CLINICAL TRIAL: NCT06697288
Title: Evaluation of the Efficacy of the UVMune 400 Fluid Sunscreen on the Face Versus Usual Photoprotection Routine on Visible and Measurable Signs of Aging
Brief Title: Evaluation of Efficacy of Anthelios Sunscreen on Face Versus Usual Routine on Signs of Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LRP23007-2223CBCL064 Anthelios
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Aging
Keywords: skin aging; Anthelios UVMUNE 400 Oil Control Fluid SPF 50+; preventive effect
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tested product group (Experimental): Volunteers using the investigational product handed over to them
  Interventions: Other: Tested product group
- Control group (Active Comparator): Volunteers using their own sun protection routine
  Interventions: Other: Control group

INTERVENTIONS:
Other: Tested product group — Apply the test product per zone at least twice a day on the face, neck (neck & nape), décolleté and back of the hand in the morning and at midday whatever the weather conditions and the activities of the day
  Arms: Tested product group
Other: Control group — Maintain their normal routine of using cosmetics (cleansers and moisturizers) and normal sun protection habits (if applicable)
  Arms: Control group

SUMMARY:
This experimental, randomized study aims at evaluating the preventative effect of a Sun Protection Factor (SPF) 50+ sunscreen (Anthelios UVMUNE 400 Fluid SPF 50+) with high Ultraviolet A (UVA) protection on clinical signs of skin aging.

DETAILED DESCRIPTION:
The study will be conducted in compliance with the protocol, current internal procedures and in the spirit of the International Council on Harmonisation (ICH) Topic E6(R2)5 ref: EMA/CHMP/ICH/135/1995, ICH Good Clinical Practice (GCP) Addendum Nov 2016 and applicable regulatory requirement.

Statistical plan: Tx represents the values observed at Time x, for each parameter and by subgroup. Quantitative variables, or those that can reasonably be treated as such, will be summarized using the minimum, maximum, measures of central tendency such as the mean and median & measures of dispersion such as the standard deviation (SD). Qualitative variables will be summarized in the form of counts and percentages.

For each parameter, a graphical representation of the means ±95% Confidence Interval (CI) will be produced to visually assess the evolution across time, by treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with signs of photo aging (Global score of at least 14)
* All skin types

Exclusion Criteria:

* Any history of significant dermatological/ophthalmological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site
* Pregnant or breastfeeding women
* Subject with known allergy to cosmetic products or to any ingredient of the sunscreen product

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Change in the dermatological assessment of skin signs on the face (Global score) | Day0; Day84; Day168; Day252; Day336
  Assessment of the skin parameters: Skin roughness [absent (0), mild (2), moderate (4), severe (6)]; Skin laxity [absent (0), mild (2), moderate (4), severe (6)]; Skin suppleness [high(0), moderate (2),low (4), absent (6)]; Skin radiance [highly radiant (0), radiant (2), normal(4), dull(6), highly dull(8)]; Pigmented spots [absent (0), visible (2), highly visible (4)]; Skin tone homogeneity [homogeneous (0), non-homogeneous (2)].

SECONDARY OUTCOMES:
Dermatological assessment of skin signs on the face - Atlas Bazin, Flament (Global score) | Day0; Day84; Day168; Day252; Day336
  Assessment of the skin parameters: Forehead wrinkles (0 - 5); Crow feet wrinkles number (1 - 4); Crow feet wrinkles deepness (1 - 6); Glabellar wrinkles (0 - 5); Glabellar fine lines (0 - 5); Underneath eye wrinkle (0 - 5); Corner mouth wrinkle (0 - 6); Nasolabial fold (0 - 5); Upper lip wrinkles (0 - 6); Neck fold (0 - 5); Neck sagging (0 - 5); Ptosis (0 - 5); Eye bags (0 - 5

CONTACTS AND LOCATIONS:
Overall Officials: Renato Moura, Principal Investigator — Centre International de Développement Pharmaceutique
Locations (1):
- CIDP, Rio de Janeiro, Brazil